CLINICAL TRIAL: NCT04913675
Title: A Phase 3 Randomized, Multi-center, Open Label Study to Assess the Efficacy, Safety, and Tolerability of Monoclonal Antibody VIR-7831 (Sotrovimab) Given Intramuscularly Versus Intravenously for the Treatment of Mild/Moderate Coronavirus Disease 2019 (COVID-19) in High-risk Non-hospitalized Patients; Safety Substudy Assessing the Safety and Tolerability of Single Ascending Dose Monoclonal Antibody VIR-7831
Brief Title: Intramuscular and Intravenous VIR-7831 (Sotrovimab) for Mild/Moderate COVID-19.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The safety sub-study was discontinued early in the context of evolving variants with increased fold changes in the in vitro half maximal inhibitory concentration (IC50) and uncertainty in the clinical relevance of these changes
Sponsor: Vir Biotechnology, Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR-7831-5008
Record Dates: First submitted 2021-05-27; First posted 2021-06-04 (Actual); Results first posted 2023-05-26 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-01

CONDITIONS: Covid19
Keywords: SARS-CoV-2; coronavirus disease 2019; COVID-19; early treatment; coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — sotrovimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Main Study - Sotrovimab 500 mg IV (Active Comparator)
  Interventions: Biological: sotrovimab
- Main Study - Sotrovimab 500 mg IM (Experimental)
  Interventions: Biological: sotrovimab
- Main Study - Sotrovimab 250 mg IM (Experimental)
  Interventions: Biological: sotrovimab
- Substudy (Cohort A) - Sotrovimab 2000 mg IV (Experimental)
  Interventions: Biological: sotrovimab
- Substudy (Optional Cohort B1) - Sotrovimab 2000 mg IV (Experimental)
  Interventions: Biological: Sotrovimab
- Substudy (Optional Cohort B2) - Sotrovimab 2000 mg IV (Experimental)
  Interventions: Biological: Sotrovimab
- Substudy (Optional Cohort C) - Sotrovimab up to 3000 mg IV (Experimental)
  Interventions: Biological: Sotrovimab

INTERVENTIONS:
Biological: sotrovimab — Sotrovimab 500 mg given by intravenous infusion over 15 min
  Arms: Main Study - Sotrovimab 500 mg IV
Biological: sotrovimab — Sotrovimab 500 mg given by intramuscular injection
  Arms: Main Study - Sotrovimab 500 mg IM
Biological: sotrovimab — Sotrovimab 250 mg given by intramuscular injection
  Arms: Main Study - Sotrovimab 250 mg IM
Biological: sotrovimab — Sotrovimab 2000 mg given by intravenous infusion over 60 min
  Arms: Substudy (Cohort A) - Sotrovimab 2000 mg IV
Biological: Sotrovimab — Sotrovimab 2000 mg given by intravenous infusion over 30 min
  Arms: Substudy (Optional Cohort B1) - Sotrovimab 2000 mg IV
Biological: Sotrovimab — Sotrovimab 2000 mg given by intravenous infusion over 15 min
  Arms: Substudy (Optional Cohort B2) - Sotrovimab 2000 mg IV
Biological: Sotrovimab — Sotrovimab up to 3000 mg given by intravenous infusion over 90 min
  Arms: Substudy (Optional Cohort C) - Sotrovimab up to 3000 mg IV

SUMMARY:
The COMET-TAIL main study evaluated efficacy, safety, and tolerability of IM sotrovimab versus IV sotrovimab in high-risk patients for the treatment of mild/moderate COVID-19. In the safety substudy, the aim was to evaluate the safety and tolerability of sotrovimab across a single ascending dose level and over different infusion times when given for the treatment of mild/moderate COVID-19 to participants at high risk of disease progression

Main study was completed successfully. The safety sub-study was discontinued early in the context of evolving variants with increased fold changes in the in vitro half maximal inhibitory concentration (IC50) and uncertainty in the clinical relevance of these changes.

ELIGIBILITY:
Inclusion Criteria:

* Main Study participant must be aged 12 years or older AND at high risk of progression of COVID-19 or > 55 years old
* Sub-Study participants must be aged 18 years or older at time of consent AND at high risk of progression of COVID-19 or ≥ 55 years old
* Participants must have a positive SARS-CoV-2 test result and oxygen saturation ≥94% on room air and have COVID-19 symptoms and be less than or equal to 7 days from onset of symptoms

Exclusion Criteria:

* Currently hospitalized or judged by the investigator as likely to require hospitalization in the next 24 hours
* Symptoms consistent with severe COVID-19
* Participants who, in the judgement of the investigator are likely to die in the next 7 days
* Known hypersensitivity to any constituent present in the investigational product

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1065 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (34):
  - Investigative Site, Anniston, Alabama
  - Investigative Site, Mesa, Arizona
  - Investigative Site, Tucson, Arizona
  - Investigative Site, Los Angeles, California
  - Investigative Site, Rolling Hills Estates, California
  - Investigative Site, Bradenton, Florida
  - Investigative Site, Doral, Florida
  - Investigative Site, Gainesville, Florida
  - Investigative Site, Hialeah, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, North Miami Beach, Florida
  - Investigative Site, Ormond Beach, Florida
  - Investigative Site, Palmetto Bay, Florida
  - Investigative Sites, Pembroke Pines, Florida
  - Investigative Site, Pompano Beach, Florida
  - Investigative Site, Tampa, Florida
  - Investigative Site, Atlanta, Georgia
  - Investigative Site, Idaho Falls, Idaho
  - Investigative Site, Mishawaka, Indiana
  - Investigative Site, Sterling Heights, Michigan
  - Investigative Site, Las Vegas, Nevada
  - Investigative Site, The Bronx, New York
  - Investigative Site, High Point, North Carolina
  - Investigative Site, Mount Airy, North Carolina
  - Investigative Site, Columbus, Ohio
  - Investigative Site, Smithfield, Pennsylvania
  - Investigative Site, Baytown, Texas
  - Investigative Site, Forney, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, Laredo, Texas
  - Investigative Site, Mesquite, Texas
  - Investigative Site, Pharr, Texas
  - Investigative Site, Kirkland, Washington
  - Investigative Site, Seattle, Washington
- Investigative Site, Limoges, Haute-Vienna, France
- Investigative Site, Kyiv, Ukraine

REFERENCES:
- [Derived] Shapiro AE, Sarkis E, Acloque J, Free A, Gonzalez-Rojas Y, Hussain R, Juarez E, Moya J, Parikh N, Inman D, Cebrik D, Nader A, Noormohamed N, Wang Q, Skingsley A, Austin D, Peppercorn A, Agostini ML, Parra S, Chow S, Mogalian E, Pang PS, Hong DK, Sager JE, Yeh WW, Alexander EL, Gaffney LA, Kohli A. Intramuscular vs Intravenous SARS-CoV-2 Neutralizing Antibody Sotrovimab for Treatment of COVID-19 (COMET-TAIL): A Randomized Noninferiority Clinical Trial. Open Forum Infect Dis. 2023 Jul 14;10(8):ofad354. doi: 10.1093/ofid/ofad354. eCollection 2023 Aug. PMID 37577112
- [Derived] Moya J, Temech M, Parra S, Juarez E, Hernandez-Loy R, Gutierrez JCM, Diaz J, Hussain R, Segal S, Xu C, Skingsley A, Schnell G, El-Zailik A, Sager JE, Aldinger M, Alexander EL, Acloque G. Safety, Virology, Pharmacokinetics, and Clinical Experience of High-Dose Intravenous Sotrovimab for the Treatment of Mild to Moderate COVID-19: An Open-Label Clinical Trial. Open Forum Infect Dis. 2023 Jul 10;10(7):ofad344. doi: 10.1093/ofid/ofad344. eCollection 2023 Jul. PMID 37520411
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consists of Main study and Safety sub-study. Main study was completed successfully. The safety sub-study was discontinued early in the context of evolving variants with increased fold changes in the in vitro half maximal inhibitory concentration (IC50) and uncertainty in the clinical relevance of these changes.
Pre-assignment Details: A total of 1065 participants were enrolled in this study (983 in main study and 82 in safety sub-study), of which 10 participants from main study and 1 from safety sub-study did not receive study intervention. Hence, a total of 973 from main study and 81 from safety sub-study were exposed to study intervention constituting the Safety Populations.
Groups:
- Main Study: Sotrovimab 500 mg IV: Participants received a single dose of sotrovimab 500 milligram (mg), intravenous (IV) infusion over 15 minutes on Day 1.
- Main Study: Sotrovimab 500 mg IM: Participants received a single dose of sotrovimab 500 mg, IM dose as 2*4 milliliter (mL) injections in each dorsogluteal muscle on Day 1.
- Main Study: Sotrovimab 250 mg IM: Participants received a single dose of sotrovimab 250 mg, intramuscular (IM) dose either as a single 250 mg (4 mL) injection in the dorsogluteal muscle or as 2*2 mL injections in each deltoid muscle on Day 1.
- Safety Sub-study: Sotrovimab (2000 mg IV): Participants received a single dose of sotrovimab 2000 mg, IV infusion over 60 minutes.
Period: Main Study (Up to Week 36)
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM | Safety Sub-study: Sotrovimab (2000 mg IV)
Started | 393 | 385 | 195 | 0
Completed | 356 | 341 | 176 | 0
Not Completed | 37 | 44 | 19 | 0
Not completed — Death | 0 | 2 | 2 | 0
Not completed — Lost to Follow-up | 12 | 8 | 4 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 25 | 33 | 12 | 0
Period: Safety Sub-study (Up to Week 36)
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM | Safety Sub-study: Sotrovimab (2000 mg IV)
Started | 0 | 0 | 0 | 81
Completed | 0 | 0 | 0 | 80
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for Safety Population for Main Study and Safety Sub-study.
Groups:
- Main Study: Sotrovimab 500 mg IV: Participants received a single dose of sotrovimab 500 milligram (mg), IV infusion over 15 minutes on Day 1.
- Main Study: Sotrovimab 250 mg IM: Participants received a single dose of sotrovimab 250 mg, IM dose either as a single 250 mg (4 mL) injection in the dorsogluteal muscle or as 2*2 mL injections in each deltoid muscle on Day 1.
- Total: Total of all reporting groups
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM | Safety Sub-study: Sotrovimab (2000 mg IV) | Total
Number analyzed (Participants) | 393 | 385 | 195 | 81 | 1054
Age, Customized [Count of Participants; unit: Participants]
  12-17 years | 2 | 0 | 1 | 0 | 3
  18-64 years | 291 | 289 | 163 | 66 | 809
  >=65 years | 100 | 96 | 31 | 15 | 242
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 197 | 113 | 47 | 581
  Male | 169 | 188 | 82 | 34 | 473
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central/South Asian Heritage | 1 | 2 | 0 | 0 | 3
  Asian - South East Asian Heritage | 0 | 1 | 0 | 0 | 1
  Black or African American | 17 | 19 | 8 | 4 | 48
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  White - Arabic/North African Heritage | 10 | 21 | 8 | 0 | 39
  White - White/Caucasian/European | 362 | 336 | 176 | 77 | 951
  Mixed Race | 1 | 2 | 1 | 0 | 4
  Unknown | 0 | 3 | 1 | 0 | 4
  Missing | 1 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Percentage of Participants Who Had Progression of Coronavirus Disease 2019 (COVID-19) Through Day 29 by Hospitalization >24 Hours or Death Due to Any Cause (Weekly and Daily Imputation)
Description: Progression of COVID-19 through Day 29 as defined by hospitalization >24 hours for acute management of illness due to any cause or death. Percentage values are rounded off.
Time Frame: Up to Day 29
Population: Primary Analysis Population consisted of all randomized participants excluding participants who were randomized under Protocol Amendment Version 1 and were immunocompetent and fully vaccinated at randomization and participants who did not meet key eligibility criteria. The statistical analysis was performed only for 500 mg IV versus 500 mg IM dose. It was not planned for 250 mg IM dose per statistical analysis plan.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 378 | 376 | 183
Percentage of participants | 1.3 | 2.7 | 5.5
Statistical Analysis 1: Comparison: Main Study: Sotrovimab 500 mg IV vs Main Study: Sotrovimab 500 mg IM; Test type: Non-Inferiority — This outcome measure was analyzed using a hypothetical estimand and assessing non-inferiority of 500 mg IM dose versus 500 mg IV using a non-inferiority margin of 3.5 percent (%) on the risk difference scale. A post-hoc weekly imputation algorithm imputes the missing outcome iteratively for each week, where missing outcomes at Day 8, 15, 22, 29 are imputed; Risk Difference (RD) = 1.06, 95% CI 2-sided [-1.15 to 3.26] — Analysis was performed using a binomial regression model with identity link function and with treatment (Sotrovimab 500mg IM, 500mg IV), age (<65, =>65 years old) and gender (male, female) as covariates
Statistical Analysis 2: Comparison: Main Study: Sotrovimab 500 mg IV vs Main Study: Sotrovimab 500 mg IM; Test type: Non-Inferiority — This outcome measure was analyzed using a hypothetical estimand and assessing non-inferiority of 500 mg IM vs 500 mg IV using a non-inferiority margin of 3.5 percent (%) on the risk difference scale. A pre-specified daily imputation algorithm imputed the missing outcome iteratively for each study day starting with Day 2 and ending at Day 29; Risk Difference (RD) = 1.16, 95% CI 2-sided [-1.23 to 3.56] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Safety Sub-study: Number of Participants With Non-Serious Adverse Events (Non-SAE) and Serious Adverse Events (SAEs) Through Day 8
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any serious adverse event that, at any dose: results in death; is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or any other situation according to medical or scientific judgement. Adverse events which were not Serious were considered as Non-Serious adverse events.
Time Frame: Up to Day 8
Population: Safety Population consisted of all enrolled participants who were exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 81
Participants
  Non-SAE | 0
  SAE | 0

3. Primary Outcome: Safety Sub-study: Number of Participants With Infusion-related Reaction Including Hypersensitivity Through Day 8
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Adverse events of special interest (AESI) included infusion-related reaction including hypersensitivity. Data for number of participants with infusion-related reaction including hypersensitivity has been presented.
Time Frame: Up to Day 8
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 81
Participants | 0

4. Primary Outcome: Safety Sub-study: Number of Participants With Any Disease Related Events Through Day 8
Description: AEs related to expected progression, signs, or symptoms of COVID-19, unless more severe than expected for the participant's current clinical status and medical history, were reported as a disease related events.
Time Frame: Up to Day 8
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 81
Participants | 2

5. Secondary Outcome: Main Study: Number of Participants With Common Non-Serious Adverse Events (Non-SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Data for Common (>=1%) non-SAEs are presented.
Time Frame: Up to Week 12
Population: Safety Population consisted of all randomized participants who were exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 393 | 385 | 195
Participants | 8 | 5 | 12

6. Secondary Outcome: Main Study: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE is defined as any serious adverse event that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, significant medical events that may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed before.
Time Frame: Up to Week 36
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 393 | 385 | 195
Participants | 3 | 7 | 3

7. Secondary Outcome: Main Study: Number of Participants With Any Infusion- or Injection-related Reaction Including Hypersensitivity
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. AESI included infusion- or injection-related reaction including hypersensitivity. Data for number of participants with any infusion- or injection-related reaction including hypersensitivity has been presented.
Time Frame: Up to Week 36
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 393 | 385 | 195
Participants | 2 | 1 | 1

8. Secondary Outcome: Main Study: Number of Participants With Any Local Site Reaction by Maximum Severity After IM Administration
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. AESIs included any solicited local site reactions. AESI were graded according to the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials 2007, Food and Drug Administration, where Grade 1=Mild toxicity; Grade 2=Moderate toxicity; Grade 3=Severe toxicity; and Grade 4= Potentially life-threatening toxicity. Higher Grade indicates higher severity. Data for any worst case post-Baseline has been presented.
Time Frame: Up to Week 36
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 385 | 195
Participants
  Grade 1 | 39 | 22
  Grade 2 | 7 | 2
  Grade 3 | 1 | 0
  Grade 4 | 0 | 0

9. Secondary Outcome: Main Study: Number of Participants With Any Disease Related Events
Description: as for outcome 4
Time Frame: Up to Week 36
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 393 | 385 | 195
Participants | 18 | 16 | 20

10. Secondary Outcome: Safety Sub-study: Number of Participants With Non-SAEs Through Week 12
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Adverse events which were no serious, were considered as non-SAEs.
Time Frame: Up to Week 12
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 81
Participants | 0

11. Secondary Outcome: Safety Sub-study: Number of Participants With SAEs Through Week 36
Description: An SAE is defined as any serious adverse event that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or any other situation according to medical or scientific judgement.
Time Frame: Up to Week 36
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 81
Participants | 1

12. Secondary Outcome: Safety Sub-study: Number of Participants With Any Infusion-related Reaction Including Hypersensitivity Through Week 12
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. AESI is infusion-related reaction including hypersensitivity.
Time Frame: Up to Week 12
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 81
Participants | 0

13. Secondary Outcome: Safety Sub-study: Number of Participants With Any Disease Related Events Through Week 12
Description: as for outcome 4
Time Frame: Up to Week 12
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 81
Participants | 4

14. Secondary Outcome: Main Study: Number of Participants With Treatment-emergent Positive Anti-drug Antibody
Description: Serum samples were collected for the determination of anti-drug antibodies (ADA) using a validated electrochemiluminescent (ECL) immunoassay. The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for specificity using the confirmation assay. Samples that confirmed positive in the confirmation assay were reported as 'positive'. Confirmed positive ADA samples were further characterized in the titration assay to quasi-quantitate the amount of ADA in the sample.
Time Frame: Up to Week 24
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 393 | 385 | 195
Participants | 25 | 51 | 26

15. Secondary Outcome: Main Study: Titers of Anti-drug Antibodies Against Sotrovimab
Description: Confirmed positive ADA samples were further analyzed to obtain the titer of the antibodies. Titer is defined as the reciprocal of the highest dilution that yield results at or above the plate-based titer cut point x MRD. Titer Median and range from treatment emergent and unaffected are described below. Immunogenicity results were categorized as treatment- induced, treatment-boosted, and treatment-unaffected. Treatment-induced=those who are ADA negative or missing data at baseline and who have at least one post-dose ADA positive sample; Treatment boosted=those who are ADA positive at baseline and have a >4*Baseline titer; Treatment unaffected=those who are positive at baseline and post-Baseline titer <=4*Baseline titer or all post- Baseline negative. Treatment emergent = treatment induced or treatment boosted
Time Frame: Up to Week 24
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Titers
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 45 | 60 | 31
Titers
  Treatment-induced: number analyzed (Participants) | 24 | 50 | 26
  Treatment-induced | 80.0 [40 to 40960] | 80.0 [40 to 5120] | 80.0 [40 to 20480]
  Treatment-boosted: number analyzed (Participants) | 0 | 0 | 0
  Treatment-unaffected: number analyzed (Participants) | 21 | 10 | 5
  Treatment-unaffected | 40.0 [40 to 1280] | 60.0 [40 to 640] | 40.0 [40 to 160]

16. Secondary Outcome: Safety Sub-study: Number of Participants With Treatment-emergent Positive Anti-drug Antibody Through Week 24
Description: as for outcome 14
Time Frame: Up to Week 24
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 81
Participants | 3

17. Secondary Outcome: Safety Sub-study: Titers of Anti-drug Antibodies Against Sotrovimab Through Week 24
Description: as for outcome 15
Time Frame: Up to Week 24
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Titers
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 81
Titers
  Treatment-induced: number analyzed (Participants) | 3
  Treatment-induced | 160.0 [40 to 320]
  Treatment-boosted: number analyzed (Participants) | 0
  Treatment-unaffected ADA: number analyzed (Participants) | 6
  Treatment-unaffected ADA | 160.0 [40 to 320]

18. Secondary Outcome: Safety Sub-study: Number of Participants With Positive Neutralizing Antibodies
Description: Blood samples were collected for the determination of positive neutralizing antibodies. A neutralizing antibody assay was performed. Neutralizing antibody test was only carried out for participants who have had a positive confirmatory binding antibody test result at visit. A participant was considered positive if they had at least one positive post-Baseline neutralizing antibody result.
Time Frame: Up to Week 24
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 9
Participants | 0

19. Secondary Outcome: Main Study: Percentage of Participants Who Had Progression of COVID-19 Through Day 29 by Emergency Room Visit or Hospitalization or Death (Weekly Imputation)
Description: Progression of COVID-19 through Day 29 as defined by visit to a hospital emergency room for management of illness or hospitalization for acute management of illness for any duration and for any cause or death. Percentage values are rounded off.
Time Frame: Up to Day 29
Population: Primary Analysis Population. The statistical analysis was performed only for 500 mg IV versus 500 mg IM dose. It was not planned for 250 mg IM dose per statistical analysis plan.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 378 | 376 | 183
Percentage of participants | 2.4 | 3.2 | 6.0
Statistical Analysis 1: Comparison: Main Study: Sotrovimab 500 mg IV vs Main Study: Sotrovimab 500 mg IM; Test type: Non-Inferiority — This outcome measure was analyzed using a hypothetical estimand and assessing non-inferiority of IM dose versus IV using a non-inferiority margin of 3.5% on the risk difference scale. Weekly imputation algorithm imputes the missing outcome iteratively for each week, where missing outcomes at Day 8, 15, 22, 29 are imputed; Risk Difference (RD) = 0.86, 95% CI 2-sided [-1.56 to 3.28] — Post-hoc analysis was performed using a binomial regression model with identify link function and with treatment (Sotrovimab 500 mg IM, 500 mg IV), age (<65, >-65 years old), and sex (male, female) as covariates

20. Secondary Outcome: Main Study: Percentage of Participants Who Progress to Develop Severe and/or Critical Respiratory COVID-19 by Visit
Description: Participants were defined as progressing to develop severe respiratory COVID-19 if they required supplemental oxygen either by nasal cannula, face mask, high-flow oxygen devices, or non-invasive ventilation. Participants were defined as progressing to develop critical respiratory COVID-19 if they required invasive mechanical ventilation or extracorporeal membrane oxygenation. Percentage values are rounded off.
Time Frame: Day 8, Day 15, Day 22, and Day 29
Population: Intent-to-Treat (ITT) Population consisted of all randomized participants excluding participants who were randomized under Protocol Amendment Version 1 and were immunocompetent and fully vaccinated at randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 385 | 383 | 185
Percentage of participants
  Day 8 | 0.3 | 1.0 | 3.8
  Day 15 | 0.3 | 1.3 | 4.3
  Day 22 | 0.3 | 1.6 | 4.3
  Day 29 | 0.3 | 1.6 | 4.3

21. Secondary Outcome: Main Study: Mean Area Under the Curve (AUC) of Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Viral Load From Day 1 to Day 8
Description: AUC of SARS-CoV-2 viral load was measured by Quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) from Day 1 to Day 8 in nasopharyngeal swab samples.
Time Frame: Day 1 to Day 8
Population: Virology Population consisted of all participants in the ITT Population with a central laboratory confirmed quantifiable Baseline nasopharyngeal swab at Day 1. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*log10 copies/mL
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 287 | 278 | 136
Day*log10 copies/mL | 25.42 (34.144) | 25.56 (36.936) | 25.46 (37.899)

22. Secondary Outcome: Main Study: Mean AUC of SARS-CoV-2 Viral Load From Day 1 to Day 8 After Administration of Sotrovimab 500 mg IV and IM
Description: AUC of SARS-CoV-2 viral load was measured by qRT-PCR from Day 1 to Day 8 in nasopharyngeal swab samples. Least squares geometric mean and 90 percent (%) confidence interval has been presented.
Time Frame: Day 1 to Day 8
Population: Virology Population. Only those participants with data available at the specified time points were analyzed. The statistical analysis was performed only for 500 mg IV versus 500 mg IM dose. It was not planned for 250 mg IM dose per statistical analysis plan.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Day*log10 copies/mL
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM
Number analyzed (Participants) | 287 | 278
Day*log10 copies/mL | 25.03 [24.45 to 25.63] | 25.96 [25.35 to 26.59]
Statistical Analysis 1: Comparison: Main Study: Sotrovimab 500 mg IV vs Main Study: Sotrovimab 500 mg IM; Test type: Equivalence — IM dose was assessed for equivalence to IV based on the two-sided 90% confidence interval for the treatment ratio falling within equivalence bounds of 0.5 to 2.0; Ratio of least square(LS) geometric mean = 1.04, 90% CI 2-sided [1.00 to 1.07] — LS geometric mean was calculated for 500mg IV versus IM by using an Analysis of Covariance (ANCOVA) Model with treatment group (sotrovimab 500mg IM, 500mg IV), age (<65, =>65 years old), gender (male, female) and Baseline viral load as covariates

23. Secondary Outcome: Main Study: Change From Baseline in Viral Load as Measured by qRT-PCR at Day 8
Description: Viral load was based on nasopharyngeal swab samples and was measured by qRT-PCR. Baseline was defined as the latest non-missing value prior to dosing (or latest value on or prior to nominal Day 1 for participants that were not dosed). Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and at Day 8
Population: Virology Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 279 | 271 | 132
Log10 copies/mL | -2.979 (1.6965) | -2.752 (1.7594) | -2.488 (1.6628)

24. Secondary Outcome: Main Study: Percentage of Participants With Persistently High SARS-CoV-2 Viral Load at Day 8
Description: Percentage of participants with a persistently high viral load were categorized as >=4.1 log10 copies/mL and <4.1 log10 copies/mL. Percentage of participants with a persistently high SARS-CoV-2 viral load at Day 8 was assessed via qRT-PCR in nasopharyngeal swab samples. Percentage values are rounded off.
Time Frame: At Day 8
Population: Virology Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 279 | 271 | 132
Percentage of participants
  >=4.1 log 10 copies/mL | 13 | 12 | 17
  <4.1 log 10 copies/mL | 87 | 88 | 83

25. Secondary Outcome: Main Study: Serum Concentration of Sotrovimab After Intravenous Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of Sotrovimab.
Time Frame: Day 1: Pre-dose, Day 8, Day 15, Day 29, Week 12, Week 20 and Week 24
Population: Pharmacokinetic Population consisted of all participants in the Safety Population who had at least 1 non-missing PK assessment (non-quantifiable values were considered as non-missing values). Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per mL
Arm/Group | Main Study: Sotrovimab 500 mg IV
Number analyzed (Participants) | 393
Microgram per mL
  Day 1: Pre-dose: number analyzed (Participants) | 363
  Day 1: Pre-dose | NA (NA) — NA indicates that, data was not available as all concentration values were below the lower limit of quantification.
  Day 8: number analyzed (Participants) | 337
  Day 8 | 53.67 (54.21)
  Day 15: number analyzed (Participants) | 338
  Day 15 | 44.62 (51.54)
  Day 29: number analyzed (Participants) | 356
  Day 29 | 33.89 (72.61)
  Week 12: number analyzed (Participants) | 353
  Week 12 | 19.10 (55.20)
  Week 20: number analyzed (Participants) | 325
  Week 20 | 9.96 (53.24)
  Week 24: number analyzed (Participants) | 344
  Week 24 | 7.66 (56.73)

26. Secondary Outcome: Main Study: Serum Concentration of Sotrovimab After Intramuscular Administration
Description: Blood samples were collected at indicated time points for PK analysis of Sotrovimab.
Time Frame: Day 1: Pre-dose, Day 8, Day 15, Day 29, Week 12, Week 20 and Week 24
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per mL
Arm/Group | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM
Number analyzed (Participants) | 385 | 195
Microgram per mL
  Day 1: Pre-dose: number analyzed (Participants) | 365 | 187
  Day 1: Pre-dose | NA (NA) — NA indicates that, data was not available as all concentration values were below the lower limit of quantification. | NA (NA) — NA indicates that, data was not available as all concentration values were below the lower limit of quantification.
  Day 8: number analyzed (Participants) | 339 | 166
  Day 8 | 20.50 (88.70) | 10.93 (92.47)
  Day 15: number analyzed (Participants) | 344 | 166
  Day 15 | 20.60 (84.01) | 10.90 (77.68)
  Day 29: number analyzed (Participants) | 355 | 174
  Day 29 | 18.92 (77.00) | 10.20 (61.80)
  Week 12: number analyzed (Participants) | 333 | 171
  Week 12 | 11.15 (64.01) | 6.15 (54.22)
  Week 20: number analyzed (Participants) | 315 | 167
  Week 20 | 5.83 (65.44) | 3.19 (57.05)
  Week 24: number analyzed (Participants) | 315 | 168
  Week 24 | 4.48 (71.57) | 2.34 (62.49)

27. Secondary Outcome: Safety Sub-study: Serum Concentration of Sotrovimab After Intravenous Administration
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of Sotrovimab.
Time Frame: Day 1: Pre-dose and end of infusion; Days 3, 5, 8, 15, 29 post-dose, Weeks 12, 20 and 24 post-dose
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per mL
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 81
Microgram per mL
  Day 1, Pre-dose: number analyzed (Participants) | 62
  Day 1, Pre-dose | NA (NA) — NA indicates that, data was not available as all concentration values were below the lower limit of quantification.
  Day 1, End of Infusion: number analyzed (Participants) | 51
  Day 1, End of Infusion | 709.18 (40.19)
  Day 3: number analyzed (Participants) | 78
  Day 3 | 428.75 (37.94)
  Day 5 | 343.51 (35.31)
  Day 8: number analyzed (Participants) | 80
  Day 8 | 289.16 (36.24)
  Day 15: number analyzed (Participants) | 80
  Day 15 | 239.79 (35.37)
  Day 29: number analyzed (Participants) | 80
  Day 29 | 203.44 (35.51)
  Week 12: number analyzed (Participants) | 80
  Week 12 | 94.80 (33.55)
  Week 20: number analyzed (Participants) | 79
  Week 20 | 52.96 (39.66)
  Week 24: number analyzed (Participants) | 80
  Week 24 | 40.82 (37.08)

28. Secondary Outcome: Safety Sub-study: Area Under the Serum Concentration-time Curve From Days 1 to 29 of After Intravenous Administration (AUCD1-29) of Sotrovimab
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of Sotrovimab. Pharmacokinetic analysis of sotrovimab was conducted using non-compartmental method.
Time Frame: Day 1: Pre-dose and end of infusion; Days 3, 5, 8, 15, 29 post-dose
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/mL
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 80
day*µg/mL | 7493.9 (34.68)

29. Secondary Outcome: Safety Sub-study: Maximum Serum Concentration of Sotrovimab After Intravenous Administration (Cmax)
Description: as for outcome 28
Time Frame: Day 1: Pre-dose and end of infusion; Days 3, 5, 8, 15, 29 post-dose, Weeks 12, 20 and 24 post-dose
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 53
µg/mL | 732.5 (42.23)

30. Secondary Outcome: Safety Sub-study: Apparent Volume of Distribution at Steady State of Sotrovimab After Intravenous Administration (Vss)
Description: as for outcome 28
Time Frame: Day 1: Pre-dose and end of infusion; Days 3, 5, 8, 15, 29 post-dose, Weeks 12, 20 and 24 post-dose
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 67
Liter | 6.81 (37.72)

31. Secondary Outcome: Safety Sub-study: Area Under the Serum Concentration-Time Curve Extrapolated From Zero to Infinity of Sotrovimab After Intravenous Administration (AUC[0-inf])
Description: as for outcome 28
Time Frame: Day 1: Pre-dose and end of infusion; Days 3, 5, 8, 15, 29 post-dose, Weeks 12, 20 and 24 post-dose
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/mL
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 67
day*µg/mL | 23992.5 (34.90)

32. Secondary Outcome: Safety Sub-study: Terminal Elimination Half-life of Sotrovimab After Intravenous Administration (t1/2)
Description: as for outcome 28
Time Frame: Day 1: Pre-dose and end of infusion; Days 3, 5, 8, 15, 29 post-dose, Weeks 12, 20 and 24 post-dose
Population: as for outcome 25
Measure: Median (Full Range); unit: Day
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 67
Day | 59.432 [45.36 to 72.87]

33. Secondary Outcome: Safety Sub-study: Apparent Volume of Distribution During the Elimination Phase of Sotrovimab After Intravenous Administration (Vz)
Description: as for outcome 28
Time Frame: Day 1: Pre-dose and end of infusion; Days 3, 5, 8, 15, 29 post-dose, Weeks 12, 20 and 24 post-dose
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 67
Liter | 7.05 (37.66)

34. Secondary Outcome: Safety Sub-study: Clearance of Sotrovimab After Intravenous Administration (CL)
Description: as for outcome 28
Time Frame: Day 1: Pre-dose and end of infusion; Days 3, 5, 8, 15, 29 post-dose, Weeks 12, 20 and 24 post-dose
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 67
mL/day | 83.4 (34.90)

35. Secondary Outcome: Safety Sub-study: Time to Reach Maximum Serum Concentration of Sotrovimab After Intravenous Administration (Tmax)
Description: as for outcome 28
Time Frame: Day 1: Pre-dose and end of infusion; Days 3, 5, 8, 15, 29 post-dose, Weeks 12, 20 and 24 post-dose
Population: as for outcome 25
Measure: Median (Full Range); unit: Day
Arm/Group | Safety Sub-study: Sotrovimab (2000 mg IV)
Number analyzed (Participants) | 53
Day | 0.044 [0.04 to 4.07]

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs were collected up to Week 36 and non-serious AEs were collected up to Week 12 for main study and safety sub-study
Description: All-cause mortality, non-SAE and SAEs were collected for main study and safety sub-study using Safety Population
Arm/Group | Main Study: Sotrovimab 500 mg IV | Main Study: Sotrovimab 500 mg IM | Main Study: Sotrovimab 250 mg IM | Safety Sub-study: Sotrovimab (2000 mg IV)
All-Cause Mortality (participants affected / at risk) | 0/393 | 2/385 | 2/195 | 0/81
Serious Adverse Events (participants affected / at risk) | 3/393 | 7/385 | 3/195 | 1/81
Other Adverse Events (participants affected / at risk) | 8/393 | 5/385 | 12/195 | 0/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: Sotrovimab 500 mg IV (N=393) | Main Study: Sotrovimab 500 mg IM (N=385) | Main Study: Sotrovimab 250 mg IM (N=195) | Safety Sub-study: Sotrovimab (2000 mg IV) (N=81)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial mass (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: Sotrovimab 500 mg IV (N=393) | Main Study: Sotrovimab 500 mg IM (N=385) | Main Study: Sotrovimab 250 mg IM (N=195) | Safety Sub-study: Sotrovimab (2000 mg IV) (N=81)
Activated partial thromboplastin time prolonged (Investigations) | 5 (5) | 2 (2) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The pre-specified daily imputation resulted in overly high inflation in the estimated progression rates for missing data. To reduce this bias and to account for progression history, weekly imputation was used for final conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol: Main Study (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT04913675/Prot_002.pdf
  • Study Protocol: Safety Substudy (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT04913675/Prot_003.pdf
  • Statistical Analysis Plan: Safety Substudy (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT04913675/SAP_004.pdf
  • Statistical Analysis Plan: Main Study (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT04913675/SAP_005.pdf